CLINICAL TRIAL: NCT05755594
Title: A Prospective Study on the Safety and Efficacy of Robot-assisted Pancreaticoduodenectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of University of South China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: USC-4310
Record Dates: First submitted 2023-02-23; First posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-02

CONDITIONS: Pancreatic Cancer; Common Bile Duct Diseases; Periampullary Carcinoma
Keywords: Robot-assisted pancreaticoduodenectomy; Safety and Efficacy; randomized controlled trial
MeSH Terms: conditions — Pancreatic Neoplasms; Common Bile Duct Diseases

STUDY DESIGN:
Masking Description: The way of surgery.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Robot-assisted Pancreaticoduodenectomy (Other): By performing pancreaticoduodenectomy on the subject using the latest generation Da Vinci robotic surgical system and assisted by another surgeon for the entire procedure
  Interventions: Procedure: Robot-assisted Pancreaticoduodenectomy

INTERVENTIONS:
Procedure: Robot-assisted Pancreaticoduodenectomy — By performing pancreaticoduodenectomy on the subject using the latest generation Da Vinci robotic surgical system and assisted by another surgeon for the entire procedure

SUMMARY:
Further studies are needed to investigate the prognosis and perioperative safety of patients undergoing robotic-assisted pancreaticoduodenectomy. In this study, clinical data and prognostic data of patients undergoing this procedure were prospectively collected and analyzed to explore its safety and efficacy.

DETAILED DESCRIPTION:
Perioperative clinical data and prognostic data of patients undergoing robotic-assisted pancreaticoduodenectomy were collected and analyzed to explore the safety and efficacy of this surgical approach.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Preoperative imaging suggested the presence of space occupying in the head of the pancreas, ampullary abdomen, and distal common bile duct tumor lesions to be treated with Pancreaticoduodenectomy
* No distant transfer
* No significant vascular invasion was received

Exclusion Criteria:

* With tumors of other organs
* Patients unable to tolerate anesthesia and operation due to serious abnormalities in functions of heart, lung and other important organs
* Patients found intraoperative peripheral organ metastasis combined with excision of other organs or found intraoperative radical excision could not be performed and underwent palliative drainage surgery or end the surgery
* Preoperative adjuvant therapy was given

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2031-06-01 (Estimated)

PRIMARY OUTCOMES:
Rate of long-term Survival | 3 years
  survival will be documented 3 years after surgery

SECONDARY OUTCOMES:
Unplanned re-admission rate after discharge within 30 days | 3 months
  Serious discomfort requiring re-admission within 30 days after discharge will be recorded, and the safety of the surgical method will be evaluated by this indicator
Incidence of postoperative complications | 2 months
  During hospitalization, common complications of pancreaticoduodenectomy, such as postoperative pancreatic fistula, bile leak, gastrojejunostomy leak, and delayed gastric emptying, will be recorded according to the international diagnostic criteria to evaluate the short-term safety of this surgical approach

CONTACTS AND LOCATIONS:
Overall Officials: Guodong Chen, PhD, Study Chair — The First Affiliated Hospital of University of South China

IPD SHARING:
Plan to Share IPD: No